CLINICAL TRIAL: NCT02130349
Title: IBDSL Biobank Project. Molecular Markers for Diagnosis and Therapy Response in IBD. A Prospective Population Based Biobank of Inflammatory Bowel Disease Patients in Zuid Limburg, The Netherlands.
Brief Title: IBDSL Biobank Project. Molecular Markers for Diagnosis and Therapy Response in IBD.
Acronym: IBDSL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IBDSL biobank project
Record Dates: First submitted 2014-04-24; First posted 2014-05-05 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: IBD; Crohns Disease; Ulcerative Colitis
Keywords: IBD; Crohns Disease; Ulcerative Colitis; Cohort; Biobank; Population based; IBDSL
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Biospecimen Retention: Samples With DNA — DNA Serum Plasma Stool Exhaled air Biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Crohns Disease: IBD patients diagnosed with Crohn's disease
- Ulcerative colitis: IBD patients diagnosed with ulcerative colitis
- IBD-Undefined: IBD patients with undefined IBD

SUMMARY:
The IBD South Limburg (IBDSL) project was initially designed as a prospective population based cohort study. Since 1991, all new IBD cases have been enrolled in the cohort and prospectively followed. As from 2011, the cohort is being scaled up into a population based biobank and focus expanded from epidemiology towards exploring underlying biologic mechanisms and identifying markers to predict disease course or therapy response.

Every adult IBD patient, diagnosed in and permanently residing in South Limburg (The Netherlands), is eligible to participate. The population based nature was reached via a multi-faceted approach; incident cases were prospectively identified through the participating hospitals, and missed patients were retrospectively identified using the nationwide histopathology registry. In 2011, over 3500 patients were included, which represents 93% of the IBD population in South Limburg.

The cohort includes baseline data, such as IBD phenotype, extent, location, behaviour, extra intestinal manifestations, medication, surgery, comorbidity and demographics. Data has prospectively been updated through chart review (clinical data), questionnaires (i.e. quality of life) and linkage to the authority database (vital state, residence). The biobank includes serum, plasma, DNA, faeces, biopsies and exhaled air.

We welcome new collaborations. Applications for collaboration are first to be approved by our IBD-SL committee.

DETAILED DESCRIPTION:
Background: Inflammatory Bowel Disease (IBD), encompassing Crohn's Disease (CD) and Ulcerative Colitis (UC), is a chronic disabling condition of the intestine. Most patients experience sequences of exacerbation in which quality of life is often impaired. Also society endures heavily, as IBD healthcare costs are estimated at 4.6-5.6 billion euros per year and high rates of unemployment and work disability are reported. The current incidence estimate is 256.000 Europeans per year, and yet increases.

IBD arises from complex interactions between a genetically altered intestinal immune response, environmental factors and intestinal microbiota. Disease phenotypes are heterogeneous and predicting individual disease course or therapy response is still merely possible; treatment of choice for instance remains a trial-and-error based succession of regimens. Further exploration of the underlying biologic mechanisms, and the identification and validation of non-invasive markers to predict disease course and therapy response are the foremost challenges in IBD field at this moment.

Deeply phenotyped IBD cohorts with a biobank are ideal tools for this type of research, and are warranted. Most IBD biobanks reflect hospital based populations thereby over representing severe and therapy refractory patients. However, many hypotheses require designs with a full IBD spectrum. Secondly, phenotypes are mostly ascertained retrospectively, which makes results prone for bias. As no prospective population based biobank excists, we started the population based IBD South Limburg (IBDSL) biobank project.

IBDSL: The IBDSL project was first established in 1991, when gastroenterologists started prospectively registering all IBD patients residing in South Limburg, the Netherlands. As from 2011, this cohort is being scaled up into a biobank and focus expanded from epidemiology towards exploring underlying biologic mechanisms and identifying markers to predict disease course or therapy response.

Population: Every adult IBD patient, diagnosed in South Limburg after 1991 and permanently residing in South Limburg (the Netherlands), is eligible to participate. The population based nature was reached via a multi-faceted approach; incident cases were prospectively identified through the participating hospitals, and missed patients were retrospectively identified using the nationwide histopathology registry. In 2011, over 3500 patients were included, representing >93% of the IBD population in South Limburg. Adults and partners of included patients serve as controls.

Datacollection: All eligible IBD patients will be contacted and asked to participate. Patients will be visited at home or in hospital by a research nurse. After informed consent, DNA, serum, plasma, exhaled air and stool are collected. All data will be added into a custommade web-based data management system (MACRO). All biomaterials are stored in the central biobank facility of the MUMC.

Additional information: IBDSL is a Dutch consortium comprising the gastroenterology departments of Maastricht University Medical Centre+ and the general district hospitals Orbis MC Sittard-Geleen and Atrium MC Heerlen. IBDSL is investigator initiated and has been funded by the consortium members. IBDSL has been approved by the Ethics Committee of the Maastricht University Medical Centre (METC 10-2-071, NL31636.068.10), and meets the ethical standards of the declaration of Helsinki. We welcome new collaborations. Applications for collaboration are first to be approved by our IBD-SL committee.

ELIGIBILITY:
Inclusion Criteria:

* All adult IBD patients (>18 years) residing permanently in South Limburg are eligible. IBD was diagnosed by certified gastroenterologists according to the Lennard-Jones criteria, and was proven by endoscopic and/or radiologic evidence and by histologic evidence.

Exclusion Criteria:

* <18 years,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult IBD patients (>18 years) residing permanently in South Limburg are eligible. IBD was diagnosed by certified gastroenterologists according to the Lennard-Jones criteria, and was proven by endoscopic and/or radiologic evidence and by histologic evidence.
  To capture the full South Limburg IBD population, a multifaceted approach was used. Incident cases were prospectively identified through the three hospitals. Missed patients were retrospectively identified using PALGA, the nationwide histopathology registry containing data on all endoscopic biopsies.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2011-02; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of seral, fecal, or volatile (exhaled air) biomarkers that reflect disease course and therapy response. | Disease course is monitored at baseline, and at every consequent hospital visit (at least annually) until lost-to-follow-up (death, migration out of region, withdraw). Biomaterial is collected at a (non-specified) timepoint after diagnosis.
  Primary aim of IBDSL: identify/validate markers that predict disease course and therapy response.
  Focus lies on all future potent biomarkers (not possible to specify at this timepoint) in blood, dna, faeces, exhaled air and biopsies. Identifying new biomarkers is done by a bolomic approach, in order to find a biomarker(-set) that predict specific aspects of disease course (severe or mild disease course, occurence of extra-intestinal manifestations and/or surgery) and therapy response (chance of therapy success). Validation of already identified biomarkers will be done in a hypothesis driven approach.
  Disease course and therapy response are reflected by endoscopic activity, clinical activity scores, number of flares, hospitalisations, surgeries, extra intestinal manifestations, comorbidity. These parameters are monitored at baseline, and at every consequent hospital visit (at least annually) until lost-to-follow-up (death, migration out of region, withdraw).

SECONDARY OUTCOMES:
Epidemiologic parameters | Disease course is monitored at baseline, and at every consequent hospital visit (at least annually) until lost-to-follow-up (death, migration out of region, withdrawal). Epidemiologic parameters are determined annually (since 1991)
  Secondary aim of IBDSL: Periodic analysis of epidemiologic parameters
  Epidemiology is reflected by incidence, prevalence, mortality, standardized comorbidic incidence ratios, and (environmental) assocations/risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Marieke Pierik, PhD, MD, Principal Investigator — Maastricht University Medical Center
Locations (3):
- Netherlands (3):
  - Atrium Medical Centre, Heerlen, Limburg
  - Maastricht University medical Center, Maastricht, Limburg
  - Orbis Medical Centre, Sittard, Limburg